CLINICAL TRIAL: NCT01919593
Title: The Efficacy of 2% Chlorhexidine Gluconate in 70% Alcohol Compared With 10% Povidone Iodine in Reducing Blood Culture Contamination in Pediatric Patients
Brief Title: Efficacy of 2% Chlorhexidine Gluconate in 70% Alcohol Compare 10% Povidone Iodine in Blood Culture in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Auchara Tangsathapornpong, Associate Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTU-PE-3-053/55
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Bacteremia
Keywords: Blood culture; Contamination; Chlorhexidine gluconate; Povidone iodine
MeSH Terms: conditions — Bacteremia | interventions — chlorhexidine gluconate; Ethanol; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% Chlorhexidine Gluconate (Experimental): apply 2% Chlorhexidine Gluconate in 70% Alcohol on skin before venipuncture
  Interventions: Drug: 2% chlorhexidine gluconate in 70% alcohol
- 10% povidone iodine (Active Comparator): apply 10% povidone iodine on the skin before venipuncture
  Interventions: Drug: 10%povidone iodine

INTERVENTIONS:
Drug: 2% chlorhexidine gluconate in 70% alcohol — skin preparation before venipuncture for blood culture in even month
  Other Names: Chloraprep
  Arms: 2% Chlorhexidine Gluconate
Drug: 10%povidone iodine — skin preparation before venipuncture for blood culture in odd month
  Other Names: Betadine
  Arms: 10% povidone iodine

SUMMARY:
To evaluate the efficacy of 2% chlorhexidine gluconate in 70% alcohol compared with 10% povidone iodine in reducing blood culture contamination in pediatric patients.

DETAILED DESCRIPTION:
This is a prospective study of pediatric patients between 0-15 years of age who were admitted in three pediatric wards: general pediatric ward aged <5 years, general pediatric ward aged >5 years, and pediatric intensive care unit at a tertiary-care teaching hospital. Patients who needed percutaneous blood cultures were eligible for enrollment and were classified into two groups according to antiseptic used: 10% povidone iodine in odd months and 2% chlorhexidine gluconate in 70% alcohol in even months. Blood cultures were taken primarily by ward nurses using standard technique. The blood cultures were analysed and monitored for 5 days. Isolated organisms and their antimicrobial susceptibilities were determined using standard microbiologic techniques.

Blood culture isolates were categorized into two groups including a true pathogen and a contaminant by clinical criteria combined with laboratory data. A blood culture was classified as contaminated if common skin flora such as Coagulase negative staphylococci, Corynebacterium spp., Micrococcus spp., or Bacillus spp. were isolated from one of the blood culture samples without isolation of the same organism from another potential infection site (for example, intravenous catheter), or a common skin flora was isolated in a patient with incompatible clinical features and improved without specific treatment for that organism.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 0-15 years of age who were admitted in three pediatric wards: general pediatric ward aged <5 years, general pediatric ward aged >5 years, and pediatric intensive care unit. Patients who needed percutaneous blood cultures were eligible for enrollment.

Exclusion Criteria:

* Preterm infant
* Patient who had skin infection at site of venepuncture
* Patient who had history allergy to 2% Chlorhexidine gluconate in 70% alcohol or 10% povidone-iodine

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1269 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
efficacy of 2% chlorhexidine gluconate in 70% alcohol compared with 10% povidone iodine | 5 days
  Pediatric patients who needed percutaneous blood cultures were recruited and were assigned 10% povidone iodine in odd months and 2% chlorhexidine gluconate in 70% alcohol in even months as an antiseptic for blood cultures. Blood culture isolates were categorized into two groups including a true pathogen and a contaminant by clinical criteria combined with laboratory data.

SECONDARY OUTCOMES:
safety of 2% chlorhexidine gluconate in 70% alcohol compared with 10% povidone iodine | 48 hours
  direct observe skin reaction after use both antiseptics

CONTACTS AND LOCATIONS:
Overall Officials: Auchara Tangsathapornponng, MD, Principal Investigator — Faculty of Medicine, Thammasat University
Locations (1):
- Thammasat University hospital, Klong Luang, Pathumthanii, Thailand